CLINICAL TRIAL: NCT01454076
Title: A Phase 1 Study of Oral IXAZOMIB (MLN9708) to Assess Relative Bioavailability, Food Effect, Drug-Drug Interaction With Ketoconazole, Clarithromycin or Rifampin; and Safety and Tolerability in Patients With Advanced Nonhematologic Malignancies or Lymphoma
Brief Title: Pharmacokinetics Study of Oral IXAZOMIB in Participants With Advanced Nonhematologic Malignancies or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C16009; U1111-1183-0218 (Registry Identifier: WHO)
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Results first posted 2017-11-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-06

CONDITIONS: Nonhematologic Malignancies; Lymphoma
Keywords: Cmax: maximum plasma concentration; AUC0-tlast: area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
MeSH Terms: conditions — Lymphoma | interventions — ixazomib; Ketoconazole; Rifampin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg (Experimental): Ixazomib 2.5 milligram (mg), capsule B, orally, once on Day 1 and 15 along with ketoconazole 400 mg, tablets, orally, once daily from Day 12 to 25 of Cycle 1 (28-day treatment cycle). After Cycle 1, participants will receive ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-day treatment cycle) up to a maximum of 12 cycles, until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib 2.5 mg; Drug: Ixazomib 4 mg Capsule B; Drug: Ketoconazole
- Arm 2: Ixazomib 4 mg Capsule A or B (Experimental): Ixazomib 4 mg, capsule A, orally, once on Day 1 followed by ixazomib 4 mg, capsule B once on Day 15 of Cycle 1 (28-day treatment cycle) or ixazomib 4 mg, capsule B, orally, once on Day 1 followed by ixazomib 4 mg, capsule A once on Day 15 of Cycle 1 (28-day treatment cycle). After Cycle 1, participants will receive ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-treatment cycle) up to a maximum of 12 cycles, until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib 4 mg Capsule A; Drug: Ixazomib 4 mg Capsule B
- Arm 3: Ixazomib 4 mg Fasted or Fed (Experimental): Ixazomib 4 mg, capsule B, orally, under fasted state, once on Day 1 followed by ixazomib 4 mg, capsule B, orally, under fed state, once on Day 15 of Cycle 1 (28-day treatment cycle) or ixazomib 4 mg, capsule B, orally, under fed state, once on Day 1 followed by ixazomib 4 mg, capsule B, orally, under fasted state, once on Day 15 of Cycle 1 (28-day treatment cycle). After Cycle 1, participants will receive ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-day treatment cycle) up to a maximum of 12 cycles, until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib 4 mg Capsule B
- Arm 4: Ixazomib 4 mg + Rifampin 600 mg (Experimental): Ixazomib, 4 mg, capsule B, orally, once on Day 8 along with rifampin 600 mg, capsule, orally, once daily from Day 1 to 14 of Cycle 1 (21-day treatment cycle). After Cycle 1, participants will receive ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-day treatment cycle) up to a maximum of 12 cycles, until disease progression or unacceptable toxicity.
  Interventions: Drug: Rifampin; Drug: Ixazomib 4 mg Capsule B
- Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg (Experimental): Ixazomib, 2.5 mg, capsule B, orally, once on Day 6 along with clarithromycin, 500 mg, tablet, orally, twice daily from Day 1 to 16 of Cycle 1 (21-day treatment cycle). After Cycle 1, participants will receive ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-day treatment cycle) up to a maximum of 12 cycles, until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib 2.5 mg; Drug: Ixazomib 4 mg Capsule B; Drug: Clarithromycin

INTERVENTIONS:
Drug: Ixazomib 2.5 mg — Ixazomib 2.5 mg Capsule B (Cycle 1 only)
  Arms: Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg; Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg
Drug: Ixazomib 4 mg Capsule A — Ixazomib 4 mg Capsule A (Cycle 1 only)
  Arms: Arm 2: Ixazomib 4 mg Capsule A or B
Drug: Ixazomib 4 mg Capsule B — Ixazomib 4 mg Capsule B (Cycle 2 and beyond )
  Arms: Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg; Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg
Drug: Ketoconazole — Ketoconazole 400 mg tablets (Cycle 1 only)
  Arms: Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg
Drug: Rifampin — Rifampin 600 mg capsule (Cycle 1 only)
  Arms: Arm 4: Ixazomib 4 mg + Rifampin 600 mg
Drug: Clarithromycin — Clarithromycin 500 mg tablets (Cycle 1 only)
  Arms: Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg
Drug: Ixazomib 4 mg Capsule B — Ixazomib 4 mg Capsule B (Cycle 1 and beyond)
  Arms: Arm 2: Ixazomib 4 mg Capsule A or B; Arm 3: Ixazomib 4 mg Fasted or Fed; Arm 4: Ixazomib 4 mg + Rifampin 600 mg

SUMMARY:
This is an open-label, multicenter, sequential, 5-arm, phase 1 study of oral IXAZOMIB designed to assess drug-drug interaction with ketoconazole (Arm 1), the relative bioavailability of 2 capsule formulations of IXAZOMIB (Arm 2), food effect (Arm 3), drug-drug interaction with rifampin (Arm 4), and drug-drug interaction with clarithromycin (Arm 5) in participants with advanced nonhematologic malignancies or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 years or older.
* Participants must have a diagnosis of histologically or cytologically confirmed metastatic and/or advanced solid tumor malignancy or lymphoma for which no effective standard treatment is available.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Female participants who are postmenopausal at least 1 year, or surgically sterile, or if of childbearing potential, agree to practice 2 effective methods of contraception, at the same time from the time of signing the consent form through 90 days after the last dose of study drug, or agree to practice true abstinence.
* Male participants, even if surgically sterilized, agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug or agree to practice true abstinence.
* Voluntary written informed consent.
* Clinical laboratory values as specified in protocol.
* Suitable venous access.
* Recovered (that is, less than [< ] Grade 1 toxicity or participant's baseline status) from the reversible effects of prior anticancer therapy.

Exclusion Criteria:

* Peripheral neuropathy greater than (>) Grade 2 on clinical examination.
* Systemic treatment with strong inhibitors of cytochrome P450 (CYP) 1A2, strong inhibitors of CYP3A, or strong CYP3A inducers or use of ginkgo biloba or St. John's wort within 14 days before the first dose of IXAZOMIB.
* Participant has symptomatic brain metastasis. Participants with brain metastases must: have stable neurologic status following surgery or radiation for at least 2 weeks after completion of the definitive therapy; and be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Female participants who are pregnant or lactating.
* Serious illness that could interfere with protocol completion.
* Autologous stem cell transplant within 6 months before Day 1 of Cycle 1, or prior allogeneic stem cell transplant at any time.
* Prior treatment with rituximab or other unconjugated any antibody treatment within 42 days (21 days if there is clear evidence of progressive disease or immediate treatment is mandated).
* Ongoing treatment with corticosteroids.
* Radiotherapy within 21 days before the first dose of study drug.
* Major surgery within 14 days before the first dose of study drug.
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days prior to first dose of study drug.
* Life-threatening illness unrelated to cancer.
* Known human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive, or suspected hepatitis C infection.
* Diagnosis or treatment of another malignancy within 2 years preceding first dose, or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Evidence of uncontrolled cardiovascular conditions.
* QTc > 500 milliseconds on a 12-lead electrocardiogram (ECG).
* Known gastrointestinal disease or procedure that could interfere with the oral absorption or tolerance of IXAZOMIB including difficulty swallowing capsules; diarrhea > Grade 1 despite supportive therapy.
* Participants with gastric achlorhydria (Arm 1 only).
* Participants who have used any nicotine containing products within 14 days before the first dose of study drug (Arm 1, Arm 4, and Arm 5).
* Treatment with any investigational products or systemic antineoplastic therapies within 21 days before the first dose of IXAZOMIB.
* Participants with known hypersensitivity to macrolide antibiotics (example, clarithromycin, erythromycin, azithromycin) or a history of jaundice/liver injury during prior exposure to clarithromycin (Arm 5 only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-11-10 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2016-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Dallas, Texas, United States

REFERENCES:
- [Derived] Gupta N, Hanley MJ, Venkatakrishnan K, Bessudo A, Rasco DW, Sharma S, O'Neil BH, Wang B, Liu G, Ke A, Patel C, Rowland Yeo K, Xia C, Zhang X, Esseltine DL, Nemunaitis J. Effects of Strong CYP3A Inhibition and Induction on the Pharmacokinetics of Ixazomib, an Oral Proteasome Inhibitor: Results of Drug-Drug Interaction Studies in Patients With Advanced Solid Tumors or Lymphoma and a Physiologically Based Pharmacokinetic Analysis. J Clin Pharmacol. 2018 Feb;58(2):180-192. doi: 10.1002/jcph.988. Epub 2017 Aug 11. PMID 28800141
- [Derived] Hanley MJ, Gupta N, Venkatakrishnan K, Bessudo A, Sharma S, O'Neil BH, Wang B, van de Velde H, Nemunaitis J. A Phase 1 Study to Assess the Relative Bioavailability of Two Capsule Formulations of Ixazomib, an Oral Proteasome Inhibitor, in Patients With Advanced Solid Tumors or Lymphoma. J Clin Pharmacol. 2018 Jan;58(1):114-121. doi: 10.1002/jcph.987. Epub 2017 Aug 7. PMID 28783865
- [Derived] Gupta N, Hanley MJ, Venkatakrishnan K, Wang B, Sharma S, Bessudo A, Hui AM, Nemunaitis J. The Effect of a High-Fat Meal on the Pharmacokinetics of Ixazomib, an Oral Proteasome Inhibitor, in Patients With Advanced Solid Tumors or Lymphoma. J Clin Pharmacol. 2016 Oct;56(10):1288-95. doi: 10.1002/jcph.719. Epub 2016 Mar 17. PMID 26872892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States from 10 November 2011 to 16 June 2016. An additional 1 center was activated but did not screen or enroll any participants.
Pre-assignment Details: Participants with advanced nonhematologic malignancies or lymphoma were enrolled in this 5 arm study to receive one of the following treatments in Cycle 1: ixazomib + ketoconazole; ixazomib Capsule A or B formulation; ixazomib in fasted or fed state; ixazomib + rifampin; ixazomib + clarithromycin; Cycle 2 up to Cycle 12: ixazomib alone in all arms.
Groups:
- Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg: Ixazomib 2.5 milligram (mg), capsule B, orally, once on Day 1 and 15 along with ketoconazole 400 mg, tablets, orally, once daily from Day 12 to 25 of Cycle 1 (28-day treatment cycle). After Cycle 1, participants received ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-day treatment cycle) up to a maximum of 12 cycles, until disease progression or unacceptable toxicity.
- Arm 2: Ixazomib 4 mg Capsule A or B: Ixazomib 4 mg, capsule A, orally, once on Day 1 followed by ixazomib 4 mg, capsule B once on Day 15 of Cycle 1 (28-day treatment cycle) or ixazomib 4 mg, capsule B, orally, once on Day 1 followed by ixazomib 4 mg, capsule A once on Day 15 of Cycle 1 (28-day treatment cycle). After Cycle 1, participants received ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-day treatment cycle) up to a maximum of 12 cycles, until disease progression or unacceptable toxicity.
- Arm 3: Ixazomib 4 mg Fasted or Fed: Ixazomib 4 mg, capsule B, orally, under fasted state, once on Day 1 followed by ixazomib 4 mg, capsule B, orally, under fed state, once on Day 15 of Cycle 1 (28-day treatment cycle) or ixazomib 4 mg, capsule B, orally, under fed state, once on Day 1 followed by ixazomib 4 mg, capsule B, orally, under fasted state, once on Day 15 of Cycle 1 (28-day treatment cycle). After Cycle 1, participants received ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-day treatment cycle) up to a maximum of 12 cycles, until disease progression or unacceptable toxicity.
- Arm 4: Ixazomib 4 mg + Rifampin 600 mg: Ixazomib, 4 mg, capsule B, orally, once on Day 8 along with rifampin 600 mg, capsule, orally, once daily from Day 1 to 14 of Cycle 1 (21-day treatment cycle). After Cycle 1, participants received ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-day treatment cycle) up to a maximum of 12 cycles, until disease progression or unacceptable toxicity.
- Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg: Ixazomib, 2.5 mg, capsule B, orally, once on Day 6 along with clarithromycin, 500 mg, tablet, orally, twice daily from Day 1 to 16 of Cycle 1 (21-day treatment cycle). After Cycle 1, participants received ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-day treatment cycle) up to a maximum of 12 cycles, until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg | Arm 2: Ixazomib 4 mg Capsule A or B | Arm 3: Ixazomib 4 mg Fasted or Fed | Arm 4: Ixazomib 4 mg + Rifampin 600 mg | Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg
Started | 29 | 20 | 24 | 18 | 21
Completed | 16 | 14 | 15 | 16 | 15
Not Completed | 13 | 6 | 9 | 2 | 6
Not completed — Other | 2 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 4 | 2 | 1 | 2
Not completed — Adverse Event | 8 | 2 | 7 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least one dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg | Arm 2: Ixazomib 4 mg Capsule A or B | Arm 3: Ixazomib 4 mg Fasted or Fed | Arm 4: Ixazomib 4 mg + Rifampin 600 mg | Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg | Total
Number analyzed (Participants) | 29 | 20 | 24 | 18 | 21 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (8.71) | 60.5 (13.33) | 62.3 (11.86) | 61.6 (11.33) | 60.0 (11.04) | 61.3 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 11 | 8 | 6 | 53
  Male | 12 | 9 | 13 | 10 | 15 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 3 | 1 | 4 | 16
  Not Hispanic or Latino | 26 | 15 | 21 | 17 | 17 | 96
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 4 | 0 | 0 | 11
  White | 22 | 15 | 18 | 17 | 19 | 91
  More than one race | 1 | 1 | 1 | 0 | 1 | 4
  Unknown or Not Reported | 1 | 2 | 1 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 29 | 20 | 24 | 18 | 21 | 112
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 166.6 (9.26) | 166.4 (9.64) | 170.2 (9.76) | 169.2 (10.03) | 172.6 (11.11) | 168.9 (10.00)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 77.44 (19.956) | 69.78 (13.057) | 74.09 (16.358) | 80.22 (17.183) | 81.93 (20.973) | 76.64 (18.083)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Ixazomib
Time Frame: Arm 1:Days 1, 15 and Arm 5:Day 6 pre-dose and at multiple time points(up to 264 hours[hrs])post-dose;Arm 2, 3:Days 1,15 pre-dose and at multiple time points(up to 216 hrs)post-dose;Arm 4:Day 8 pre-dose and at multiple time points(up to 168 hrs)post-dose
Population: The pharmacokinetic (PK)-evaluable population included all participants who received protocol-specified dose in Cycle 1 without dose reductions/interruptions, did not receive any excluded concomitant medication during PK sampling, and had sufficient concentration-time data to permit estimation of PK parameters by noncompartmental analysis methods.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Arm 1: Ixazomib 2.5 mg: Ixazomib 2.5 mg, capsule B, orally, once on Day 1 of Cycle 1 (28-day treatment cycle).
- Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg: Ixazomib 2.5 mg, capsule B, orally, once on Day 15 along with ketoconazole 400 mg, tablets, orally, once daily from Day 12 to 25 of Cycle 1 (28-day treatment cycle).
- Arm 2: Ixazomib 4 mg Capsule A: Ixazomib 4 mg, capsule A, orally, once on Day 1 or 15 of Cycle 1 (28-day treatment cycle).
- Arm 2: Ixazomib 4 mg Capsule B: Ixazomib 4 mg, capsule B, orally, once on Day 1 or 15 of Cycle 1 (28-day treatment cycle).
- Arm 3: Ixazomib 4 mg Fasted: Ixazomib 4 mg, capsule B, orally, under fasted conditions, once on Day 1 or 15 of Cycle 1 (28-day treatment cycle).
- Arm 3: Ixazomib 4 mg Fed: Ixazomib 4 mg, capsule B, orally, under fed conditions, once on Day 1 or 15 of Cycle 1 (28-day treatment cycle).
- Arm 4: Ixazomib 4 mg + Rifampin 600 mg: Ixazomib, 4 mg, capsule B, orally, once on Day 8 along with rifampin 600 mg, capsule, orally, once daily from Day 1 to 14 of Cycle 1 (21-day treatment cycle).
- Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg: Ixazomib, 2.5 mg, capsule B, orally, once on Day 6 along with clarithromycin, 500 mg, tablet, orally, twice daily from Day 1 to 16 of Cycle 1 (21-day treatment cycle).
Arm/Group | Arm 1: Ixazomib 2.5 mg | Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg | Arm 2: Ixazomib 4 mg Capsule A | Arm 2: Ixazomib 4 mg Capsule B | Arm 3: Ixazomib 4 mg Fasted | Arm 3: Ixazomib 4 mg Fed | Arm 4: Ixazomib 4 mg + Rifampin 600 mg | Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg
Number analyzed (Participants) | 16 | 16 | 14 | 14 | 15 | 15 | 16 | 15
nanogram per milliliter (ng/mL) | 38.975 (21.3727) | 39.250 (27.3318) | 61.866 (48.3909) | 71.949 (46.2132) | 77.001 (53.5905) | 22.752 (15.0506) | 25.706 (15.1435) | 37.245 (21.4416)

2. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Ixazomib
Time Frame: Arm 1:Days 1, 15 and Arm 5:Day 6 pre-dose and at multiple time points(up to 264 hrs)post-dose;Arm 2, 3:Days 1,15 pre-dose and at multiple time points(up to 216 hrs)post-dose;Arm 4:Day 8 pre-dose and at multiple time points(up to 168 hrs)post-dose
Population: The PK-evaluable population included all participants who received protocol-specified dose in Cycle 1 without dose reductions/interruptions, did not receive any excluded concomitant medication during PK sampling, and had sufficient concentration-time data to permit estimation of PK parameters by noncompartmental analysis methods.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)]
Arm/Group | Arm 1: Ixazomib 2.5 mg | Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg | Arm 2: Ixazomib 4 mg Capsule A | Arm 2: Ixazomib 4 mg Capsule B | Arm 3: Ixazomib 4 mg Fasted | Arm 3: Ixazomib 4 mg Fed | Arm 4: Ixazomib 4 mg + Rifampin 600 mg | Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg
Number analyzed (Participants) | 16 | 16 | 14 | 14 | 15 | 15 | 16 | 15
nanogram*hour per milliliter (ng*hr/mL)] | 551.985 (191.4490) | 1148.778 (581.4376) | 1284.079 (941.4838) | 1334.659 (1244.0951) | 1465.979 (812.0514) | 998.698 (1019.1868) | 231.527 (134.9720) | 613.112 (375.0216)

3. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Cycle 1 Day 1 up to 30 days after last dose of study drug (Arm 1 and 5: Cycle 19 Day 45; Arm 2: Cycle 7 Day 45; Arm 3: Cycle 22 Day 45; Arm 4: Cycle 25 Day 45)
Population: The safety population included all participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Groups:
- Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg: Ixazomib 2.5 mg, capsule B, orally, once on Day 1 and 15 along with ketoconazole 400 mg, tablets, orally, once daily from Day 12 to 25 of Cycle 1 (28-day treatment cycle). After Cycle 1, participants received ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-day treatment cycle) up to a maximum of 12 cycles, until disease progression or unacceptable toxicity.
- Arm 4: Ixazomib 4 mg + Rifampin 600 mg: Ixazomib, 4 mg, capsule B, orally, once on Day 8 along with rifampin 600 mg, capsule, orally, once daily from Day 1 to 14 of Cycle 1 (21-day treatment cycle). Participant received ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-day treatment cycle) up to a maximum of 12 cycles, until disease progression or unacceptable toxicity.
- Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg: Ixazomib, 2.5 mg, capsule B, orally, once on Day 6 along with clarithromycin, 500 mg, tablet, orally, twice daily from Day 1 to 16 of Cycle 1 (21-day treatment cycle). After Cycle 1, participants received ixazomib 4 mg, capsule B, orally, once daily on Days 1, 8 and 15 of each cycle (28-day treatment cycle) up to a maximum of 12 cycles (28-day treatment cycle), until disease progression or unacceptable toxicity.
Arm/Group | Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg | Arm 2: Ixazomib 4 mg Capsule A or B | Arm 3: Ixazomib 4 mg Fasted or Fed | Arm 4: Ixazomib 4 mg + Rifampin 600 mg | Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg
Number analyzed (Participants) | 29 | 20 | 24 | 18 | 21
participants
  TEAEs | 29 | 20 | 24 | 18 | 21
  SAEs | 12 | 5 | 12 | 3 | 10

4. Secondary Outcome: Number of Participants With Clinically Significant TEAEs Related to Laboratory Abnormalities
Time Frame: Cycle 1 Day 1 up to 30 days after last dose of study drug (Arm 1 and 5: Cycle 19 Day 45; Arm 2: Cycle 7 Day 45; Arm 3: Cycle 22 Day 45; Arm 4: Cycle 25 Day 45
Population: The safety population included all participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg | Arm 2: Ixazomib 4 mg Capsule A or B | Arm 3: Ixazomib 4 mg Fasted or Fed | Arm 4: Ixazomib 4 mg + Rifampin 600 mg | Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg
Number analyzed (Participants) | 29 | 20 | 24 | 18 | 21
participants
  Blood and lymphatic system disorders | 11 | 7 | 9 | 2 | 1
  Investigations | 10 | 5 | 11 | 4 | 5
  Metabolism and nutrition disorders | 22 | 12 | 13 | 6 | 6

5. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities
Time Frame: as for outcome 4
Population: The safety population included all participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg | Arm 2: Ixazomib 4 mg Capsule A or B | Arm 3: Ixazomib 4 mg Fasted or Fed | Arm 4: Ixazomib 4 mg + Rifampin 600 mg | Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg
Number analyzed (Participants) | 29 | 20 | 24 | 18 | 21
participants | 0 (0.324) | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With Best Overall Response
Description: Best overall response for a participant is best observed post-baseline disease response as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1: Complete response (CR) was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than (<) 10 millimeter [mm]). No new lesions. Partial response (PR) was defined as greater than or equal to (>=) 30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. Stable disease (SD) was defined as not qualifying for CR, PR, Progressive Disease (PD). An increase of >=20% from the nadir (or baseline, if it represents the point at which the sum of target disease was lowest) represents PD.
Time Frame: Baseline up to end of treatment (approximately 1.9 years)
Population: The response-evaluable population included participants who had measurable disease at baseline, received at least 1 dose of any study drug, and had at least 1 postbaseline response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg | Arm 2: Ixazomib 4 mg Capsule A or B | Arm 3: Ixazomib 4 mg Fasted or Fed | Arm 4: Ixazomib 4 mg + Rifampin 600 mg | Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg
Number analyzed (Participants) | 16 | 14 | 17 | 17 | 18
percentage of participants
  CR | 0 [0.0 to 20.6] | 0 [0.0 to 23.2] | 0 [0.0 to 19.5] | 0 [0.0 to 19.5] | 0 [0.0 to 4.5]
  PR | 0 [0.0 to 20.6] | 0 [0.0 to 23.2] | 6 [0.1 to 28.7] | 0 [0.0 to 19.5] | 1 [0.0 to 6.7]
  SD | 63 [35.4 to 84.8] | 50 [23.0 to 77.0] | 35 [14.2 to 61.7] | 53 [27.8 to 77.0] | 53 [27.8 to 77.0]
  PD | 38 [15.2 to 64.6] | 50 [23.0 to 77.0] | 59 [32.9 to 81.6] | 47 [23.0 to 72.2] | 47 [23.0 to 72.2]

7. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Ixazomib
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Arm 1: Ixazomib 2.5 mg | Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg | Arm 2: Ixazomib 4 mg Capsule A | Arm 2: Ixazomib 4 mg Capsule B | Arm 3: Ixazomib 4 mg Fasted | Arm 3: Ixazomib 4 mg Fed | Arm 4: Ixazomib 4 mg + Rifampin 600 mg | Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg
Number analyzed (Participants) | 16 | 16 | 14 | 14 | 15 | 15 | 16 | 15
hours | 1.090 [0.47 to 2.07] | 1.500 [0.50 to 4.17] | 1.290 [0.52 to 3.00] | 1.250 [0.50 to 7.50] | 1.020 [0.48 to 4.00] | 4.000 [1.93 to 8.03] | 1.450 [0.50 to 4.12] | 1 [0.42 to 7.18]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after first dose of study drug and no more than 30 days for a serious adverse event after last dose of study drug (Cycle 25 Day 45)
Description: At each visit, investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by investigator was recorded, irrespective of relation to study treatment.
Arm/Group | Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg | Arm 2: Ixazomib 4 mg Capsule A or B | Arm 3: Ixazomib 4 mg Fasted or Fed | Arm 4: Ixazomib 4 mg + Rifampin 600 mg | Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg
Serious Adverse Events (participants affected / at risk) | 12/29 | 5/20 | 12/24 | 3/18 | 10/21
Other Adverse Events (participants affected / at risk) | 28/29 | 20/20 | 23/24 | 18/18 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg (N=29) | Arm 2: Ixazomib 4 mg Capsule A or B (N=20) | Arm 3: Ixazomib 4 mg Fasted or Fed (N=24) | Arm 4: Ixazomib 4 mg + Rifampin 600 mg (N=18) | Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg (N=21)
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Interstitial granulomatous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Ixazomib 2.5 mg + Ketoconazole 400 mg (N=29) | Arm 2: Ixazomib 4 mg Capsule A or B (N=20) | Arm 3: Ixazomib 4 mg Fasted or Fed (N=24) | Arm 4: Ixazomib 4 mg + Rifampin 600 mg (N=18) | Arm 5: Ixazomib 2.5 mg + Clarithromycin 500 mg (N=21)
Seasonal allergy (Immune system disorders) | 2 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 1 | 1 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 1 | 1 | 1 | 1
Hot flush (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 3 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 2 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 5 | 2 | 2 | 0 | 2
Insomnia (Psychiatric disorders) | 4 | 1 | 2 | 2 | 1
Confusional state (Psychiatric disorders) | 3 | 0 | 2 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 2 | 1 | 2
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 1 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 2 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 2 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 4 | 6 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 2 | 2 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 2 | 2 | 6 | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 4 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 1 | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 0 | 2
International normalised ratio increased (Investigations) | 1 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 1 | 1
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4 | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5 | 2 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin wrinkling (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 2 | 4 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 1 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 3 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 2
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Tongue atrophy (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 13 | 7 | 6 | 4 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2 | 5 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 4 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 20 | 7 | 9 | 8 | 8
Asthenia (General disorders) | 11 | 4 | 5 | 1 | 2
Chills (General disorders) | 5 | 2 | 2 | 2 | 1
Malaise (General disorders) | 0 | 2 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 1 | 1 | 2 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Device occlusion (Product Issues) | 1 | 0 | 2 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.